CLINICAL TRIAL: NCT00994643
Title: Phase II Study of IL-2 and Rituximab Maintenance in High Risk B Cell Non-Hodgkin's Lymphoma
Brief Title: Safety and Efficacy Study of Immunotherapy With Rituximab and Interleukin-2 in Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08S.461; 2008-40 (Other: CCRRC); JT 1375 (Other: JeffTrial Number)
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: High Risk Non-Hodgkin's Lymphoma
Keywords: NHL; Non Hodgkin's Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Rituximab; Interleukin-2; aldesleukin; Interleukins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Interleukin Therapy, Monoclonal Antibody) (Experimental): Patients receive interleukin-2 SC twice weekly and rituximab IV once weekly in weeks 5-8 and 25-28. Courses repeat every 4 weeks for up to 7 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Rituximab; Biological: Interleukin-2

INTERVENTIONS:
Biological: Rituximab — Given IV
  Other Names: C2B8 Monoclonal Antibody; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Biological: Interleukin-2 — Given SC
  Other Names: Aldesleukin; IL-2; Interleukin II; Proleukin; Recombinant Human Interleukin-2; Recombinant Interleukin-2; TCGF; Interleukin

SUMMARY:
This is a study to see if maintenance therapy with low dose interleukin-2 (IL-2) and rituximab can delay or prevent recurrences in patients with high risk Non-Hodgkin's Lymphoma (NHL). IL-2 is a naturally occurring cytokine in our immune system which may enhance the activity of a known therapeutic agent rituximab, a monoclonal antibody against CD-20, in the setting of NHL.

DETAILED DESCRIPTION:
Interleukin 2 (IL-2) is a naturally circulating cytokine produced by immune cells including T cells, dendritic cells and thymic cells. IL-2 is an integral part of T cell proliferation, autoimmunity and self-tolerance. Low dose IL-2 has been studied as maintenance therapy following autologous stem cell transplantation in Non-Hodgkin's Lymphoma. One early study showed that low dose IL-2 at dose of 3 million units per m2 twice a week for one year increased the activity and absolute number of natural killer (NK) cells which are a type of cytotoxic lymphocyte that is a major component of our innate immune system. More importantly, this dose of IL-2 prolonged time to progression in 9 patients with residual disease after autologous transplant and induced sustained complete remissions in two more patients. NK cells are involved in tumor killing via antibody dependent cell cytotoxicity, release of cytotoxic granules causing direct tumor killing and expression of ligands that trigger apoptosis or programmed cell death. In that study, no changes were seen in regulatory T cells which have been recently found to exert an inhibitory effect on NK cell function and hence limit the NK cell's ability to exert an anti-tumor effect.2,5 Because both regulatory T cells and NK cells express the IL-2 receptor, higher doses of IL-2 administration (14MIU SQ thrice weekly) would expand both populations of cells which may explain the lack of benefit seen in other clinical studies. At lower doses of 3MIU SQ twice weekly used in the earlier study, we anticipate selective upregulation of NK cells without effecting regulatory T cells.

Rituximab is a monoclonal antibody against CD20 antigen that is expressed in most B cell lymphomas. It is commonly used in the treatment of B cell lymphomas either alone or in combination with other therapy. It has been used as part of initial treatment after diagnosis as well as re-treatment if lymphoma recurred. It has also been studied as maintenance therapy in relapsed or resistant follicular lymphoma showing that rituximab delayed disease progression compared to the group who did not receive maintenance rituximab.11 The mechanism of action of rituximab includes complement mediated cytotoxicity, antibody dependent cellular cytotoxicity, induction of apoptosis and sensitization of cancer cells to cytotoxic chemotherapy. Antibody dependent cellular cytotoxicity is mediated by NK cells, macrophages and monocytes.13 The purpose of this study is to determine if the combination of low dose IL-2 plus rituximab is more effective than low dose IL-2 alone after primary or salvage therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20 B cell non-Hodgkin's lymphoma
* Karnofsky performance status scores of 70 or greater (ECOG performance status 0 to 2).
* Age greater than 18.
* Eligible patients will start treatment between D+30 and D+100 from end of prior therapy
* Patients have obtained a complete remission after induction chemotherapy or salvage chemotherapy who are not candidates for autologous stem cell transplantation or at least a partial remission after autologous transplantation (Stem cell collection, if indicated, should be collected prior to starting therapy)
* International Prognostic Index (IPI)* or Follicular Lymphoma IPI (FLIPI)of 3 or more
* Adequate organ function that has been determined within 2 weeks prior to the study entry, defined as:
* Absolute neutrophil count (ANC) >/=1000/mm3, platelets >/=100,000/mm3, and hemoglobin >/=8 g/dl.
* Serum bilirubin < 1.5 times ULN and serum albumin > 2.0 g/dl.
* If female, neither pregnant (negative pregnancy test) nor breast-feeding.
* If of child bearing potential (< one year post-menopausal), must agree to practice an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, condom, diaphragm with spermicidal, cervical cap, abstinence or sterile sex partner) from the time informed consent is signed.
* No other concurrent active malignancy requiring treatment.
* Able to render informed consent and to follow protocol requirements.

Exclusion Criteria:

* CNS lymphoma
* Presence of any other medical complications which imply a survival of less than three months.
* Prior IL-2 therapy
* HIV or Viral Hepatitis
* Karnofsky performance score less than 70.
* Pregnancy or breast-feeding.
* Unable or unwilling to utilize contraception if of childbearing potential.
* Severe cardiovascular disease within 12 months including myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attach, pulmonary embolism, life threatening arrhythmias, or uncontrollable hypertension.
* Autoimmune disorders
* Concurrent immunosuppressive medications
* Concurrent systemic corticosteroids at doses greater than replacement levels
* Prior history of intolerance to rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-02-05 (Actual); Primary Completion 2014-06-25 (Actual); Study Completion 2015-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Carabasi, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Interleukin Therapy, Monoclonal Antibody)
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Interleukin Therapy, Monoclonal Antibody)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Assess the Efficacy of Combination Immunotherapy With Rituximab and Interleukin-2 in Patients With Non-Hodgkin's Lymphoma
Description: Patients were enrolled based on having obtained complete remission or at least a partial remission. Efficacy was therefore determined by the number of patients that remained in remission following treatment.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Interleukin Therapy, Monoclonal Antibody)
Number analyzed (Participants) | 11
Participants | 6

ADVERSE EVENTS:
Time Frame: Two years and three months
Arm/Group | Treatment (Interleukin Therapy, Monoclonal Antibody)
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Interleukin Therapy, Monoclonal Antibody) (N=11)
Stroke (CNS cerebrovascular ischemia) (Nervous system disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 1 (1)
Infection -Simusitis (Infections and infestations) | 1 (1)
Absolute Neutrophil Count decreased (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Interleukin Therapy, Monoclonal Antibody) (N=11)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Achiness (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
ALT (Renal and urinary disorders) | 1 (4)
ALC Decreased (Blood and lymphatic system disorders) | 1 (2)
ANC decreased (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Nervous system disorders) | 3 (4)
AST (Blood and lymphatic system disorders) | 1 (1)
Awakening to urinate (Renal and urinary disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Bleeding (Blood and lymphatic system disorders) | 1 (1)
Blood in semen (Reproductive system and breast disorders) | 1 (1)
Bone pain (General disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Bruising (Blood and lymphatic system disorders) | 1 (3)
Bumps at location of IL-2 Injection (Skin and subcutaneous tissue disorders) | 1 (1)
Change in vision (Eye disorders) | 3 (4)
Chest pain (General disorders) | 3 (4)
Chest tightness (General disorders) | 1 (1)
Chills (General disorders) | 9 (14)
Cold Virus (Immune system disorders) | 2 (2)
Confusion (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Dermatology (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dizziness (General disorders) | 3 (4)
Dry eyes (Eye disorders) | 2 (2)
Dry mouth (General disorders) | 1 (2)
Dysgeusia (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema (General disorders) | 2 (2)
Fatigue (General disorders) | 10 (14)
Fever (General disorders) | 4 (6)
Flushing (Skin and subcutaneous tissue disorders) | 1 (2)
Flu like symptoms (Immune system disorders) | 4 (4)
Foot pain (General disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Headache (General disorders) | 5 (7)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (2)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (2)
Hypergylcemia (Blood and lymphatic system disorders) | 2 (3)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Injection site redness (General disorders) | 1 (2)
Injection site reaction (General disorders) | 1 (1)
Insomnia (General disorders) | 4 (5)
Itching (General disorders) | 3 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Local injection site sore (General disorders) | 3 (3)
Lump on left side of scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Mood Swings (Nervous system disorders) | 1 (1)
Mucositis (General disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (General disorders) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Neuropathy (Nervous system disorders) | 4 (4)
Night sweats (General disorders) | 1 (1)
Numbness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 3 (5)
Pain ankle (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Peripheral Neuropathy (Nervous system disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Restless leg Syndrome (Nervous system disorders) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sexual problems (Reproductive system and breast disorders) | 1 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinus congestion (General disorders) | 3 (3)
Sinus pain (General disorders) | 2 (2)
Skin lump (Skin and subcutaneous tissue disorders) | 2 (2)
Speech Change (General disorders) | 1 (1)
Stomach pain (General disorders) | 1 (1)
Sweating (General disorders) | 2 (2)
Taste alteration (General disorders) | 1 (1)
Tearing of eyes (Eye disorders) | 2 (3)
Tremors (Nervous system disorders) | 1 (2)
Trouble sleeping (General disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Reproductive system and breast disorders) | 2 (2)
Voice changes (General disorders) | 2 (2)
Vomiting (General disorders) | 2 (2)
WBC decreased (Blood and lymphatic system disorders) | 1 (1)
Weakness (General disorders) | 2 (2)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 3 (4)
Nocturnal Wheezing (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes